CLINICAL TRIAL: NCT01648283
Title: Role of CYP2B6 Polymorphisms in Methadone Metabolism and Clearance
Brief Title: CYP2B6 Polymorphisms in Methadone Disposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201203105
Record Dates: First submitted 2012-06-06; First posted 2012-07-24 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: methadone polymorphisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methadone arm (Experimental): 1. Intravenous racemic methadone HCl, 6.0 mg bolus
  2. Oral deuterated racemic methadone HCl, 11 mg capsule (IND#58,511)
  Interventions: Drug: IV racemic methadone HCl; Drug: Oral racemic methadone HCl

INTERVENTIONS:
Drug: IV racemic methadone HCl — IV racemic Methadone HC1 6 mg
Drug: Oral racemic methadone HCl — oral d5-methadone HCl 11 mg

SUMMARY:
This research study will determine if genetic variation in CYP2B6 affects how the body metabolizes methadone.

DETAILED DESCRIPTION:
This investigation determined the influence of CYP2B6 genetic variation, specifically CYP2B6*6 polymorphism, on clinical methadone plasma concentrations, clearance, and metabolism. The hypothesis was that CYP2B6*6 heterozygotes or homozygotes would have reduced metabolism and clearance. A secondary objective was to evaluate other less common genotypic variants, when encountered. Healthy volunteers in genotype cohorts CYP2B6*1/*1, CYP2B6*1/*6 , and CYP2B6*6/*6, and also CYP2B6*4 and CYP2B6*5 carriers, received single doses of IV and oral methadone. Plasma and urine methadone and metabolite concentrations were determined by tandem mass spectrometry. The primary outcome measure was methadone metabolism, measured as plasma metabolite/patent area under the concentration-time curve ratio and metabolite formation clearance.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria:

* 18-50 yr old
* CYP2B6*1/*1, CYP2B6*1/*6 or CYP2B6*6/*6 genotype
* Good general health with no remarkable medical conditions
* BMI < 33
* Provided informed consent

Exclusion Criteria:

Subjects will not be enrolled if any of the following criteria exist:

* Known history of liver or kidney disease
* Use of prescription or non prescription medications, herbals or foods known to be metabolized by or affect CYP2B6
* Females who are pregnant or nursing
* Known history of drug or alcohol addiction (prior or present addiction or treatment for addiction)
* Direct physical access to and routine handling of addicting drugs in the regular course of duty (this is a routine exclusion from studies of drugs with addiction potential)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Schoool of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Kharasch ED, Regina KJ, Blood J, Friedel C. Methadone Pharmacogenetics: CYP2B6 Polymorphisms Determine Plasma Concentrations, Clearance, and Metabolism. Anesthesiology. 2015 Nov;123(5):1142-53. doi: 10.1097/ALN.0000000000000867. PMID 26389554
- Available data/document: Publication — https://www.ncbi.nlm.nih.gov/pubmed?term=%22Anesthesiology%22[Jour]%20AND%202015[pdat]%20AND%20Kharasch[author]%20AND%20methadone%20cyp2b6&cmd=correctspelling — Study results published Anesthesiology. 2015 Nov;123(5):1142-53. doi: 10.1097/ALN.0000000000000867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subject withdrawals following consent due to personal reasons and/or conflicts, 3 subjects not evaluable, 64 subjects evaluable and included in analysis
Groups:
- Methadone Arm: 1. Intravenous racemic methadone HCl, 6.0 mg bolus
  2. Oral deuterated racemic methadone HCl, 11 mg capsule (IND#58,511) CYP2B6 is phenotyped by the clearance oral racemic bupropion 150mg
  racemic methadone HC1: IV racemic Methadone HC1 6 mg oral d5-methadon HC1 11 mg
  Oral deuterated racemic methadone HCl,: 11 mg capsule once
Period: Overall Study
Arm/Group | Methadone Arm
Started | 78
Completed | 64
Not Completed | 14
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Population: 3 subjects with non-evaluable PK data
Arm/Group | Methadone Arm
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants] — enrollment from greater St. Louis metropolitan area
  participants
    United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Methadone Metabolism
Description: Plasma metabolite EDDP/methadone area under the concentration-time curve (AUC0-96) ratio
Time Frame: up to 96 hours
Population: Plasma EDDP/methadone AUC ratio
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- CYP2B6*1/*1: Oral R-methadone HCl
- CYP2B6*1/*6; CYP2B6*6/*6: Oral R-methadone
Arm/Group | CYP2B6*1/*1 | CYP2B6*1/*6 | CYP2B6*6/*6
Number analyzed (Participants) | 21 | 20 | 17
ratio | 0.082 (0.022) | 0.073 (0.026) | 0.054 (0.017)
Statistical Analysis 1: Comparison: CYP2B6*1/*1 vs CYP2B6*1/*6 vs CYP2B6*6/*6; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Methadone Arm
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 56/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone Arm (N=67)
Nausea (Gastrointestinal disorders) | 42 (42) — Nausea and/or vomiting
Headache (General disorders) | 15 (15) — routinely related to caffeine abstinence prior to study session
Itching (Skin and subcutaneous tissue disorders) | 26 (26)
Dizzyness (General disorders) | 26 (26)
syncope (General disorders) | 1 (1) — syncopal episodes related to postural hypotension
feeling "hyperactive" (General disorders) | 1 (1) — self reported by subject, no obvious s/s
light senstivity (General disorders) | 1 — self reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No